CLINICAL TRIAL: NCT00755326
Title: Dose Escalation Study Of Chinese Herbs In Osteoarthritis Of The Knee
Acronym: TCM-OAK
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Brian Berman, Director, Center for Integrative Medicine, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HP-00040954; U19AT003266-01 (NIH)
Record Dates: First submitted 2008-09-17; First posted 2008-09-18 (Estimated); Results first posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Osteoarthritis of the Knee
Keywords: OA
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Danazol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Huo-Luo-Xiao-Ling (Active Comparator): Active herb Huo-Luo-Xiao-Ling (HLXL) The subjects in the HLXL group received the medium dose of HLXL (10 capsules/day or 4,000mg/day) in the first 2 weeks to evaluate safety. If no adverse effects were observed, the dose was increased to 14 capsules per day (5,600 mg/day) for the subsequent 6 weeks.
  Interventions: Drug: HLXL
- Placebo (Placebo Comparator): Placebo Huo-Luo-Xiao-Ling (HLXL): Subjects in the placebo group received an equal number of placebo capsule.
  Interventions: Drug: HLXL

INTERVENTIONS:
Drug: HLXL — Two daily dosages will be investigated. Huo-Luo-Xiao-Ling (HLXL) dose (10 capsules/day or 4,000mg/day) in the first 2 weeks to evaluate safety. If no adverse effects were observed, the dose was increased to 14 capsules per day (5,600 mg/ day) for the subsequent 6 weeks.
  Other Names: Huo-Luo-Xiao-Ling (HLXL) Dan

SUMMARY:
The purpose of this study is to determine if the traditional Chinese herbal compound (Huo-Luo-Xiao-Ling Dan, or HLXL) is effective in treating OA of the knee in addition to participants current OA of the knee treatment(s) and also to determine the best dosage of HLXL that is safe and well tolerated.

DETAILED DESCRIPTION:
The specific aims of this project are:

1. To determine whether HLXL improves pain and/or function in patients with OA of the knee who continue to have symptoms despite receiving standard analgesic and/or anti-inflammatory treatment,
2. To identify an optimal dosage of HLXL, among two dosages, as determined by pain relief and/or functional improvement, in a dose-escalation, placebo-controlled double-blind randomized phase II clinical trial, in conjunction with indicia of safety and tolerability in patients with OA of the knee who are receiving standard analgesic and/or anti-inflammatory treatment,
3. To explore mechanisms of action of HLXL, correlating changes in biological markers of suppression of systemic inflammation with changes in clinical response

ELIGIBILITY:
Inclusion Criteria:

* Age 40 years or above
* Diagnosis of OA of the knee of at least 6 months duration fulfilling American College of Rheumatology criteria
* Pain in at least one knee of at least moderate severity (Likert scale [none, mild, moderate, severe, extreme] or VAS pain score of at least 40 [0-100]) on most (at least 15) days of the previous 1 month
* Taking analgesic or nonsteroidal anti-inflammatory agents for control of pain
* Documented radiographic changes of osteoarthritis of the knee (Kellgren-Lawrence grade greater than or equal to 2 at the time of screening)
* Stable on arthritis medications for previous 1 month
* Willingness and ability, with help of a caregiver if necessary, to comply with treatment and follow-up procedures
* Use of effective contraception if woman of childbearing potential
* Signed consent statement

Exclusion Criteria:

* Intra-articular (IA) corticosteroid injection of either knee within a 3 month interval immediately prior to baseline screening
* IA hyaluronates in either knee within the past 6 months
* Tidal lavage or arthroscopy of either knee within the past 12 months
* Medical condition, in the judgment of the examiner and/or study investigators, that may preclude safe participation in protocol or prevents completion of the study, such as: uncontrolled angina and/or congestive heart failure, severe chronic obstructive pulmonary disease, active treatment for cancer, major psychiatric disease, other severe systemic disease, or significant abnormalities on screening physical examination and laboratory tests that reveal clinically important abnormalities of hematological, cardiac, pulmonary, metabolic, renal, hepatic, gastrointestinal or other systems
* Use of any constituent herb in HLXL within the past 3 months
* Current use of Chinese herbs for arthritis
* Use of oral prednisone in the past 30 days
* Current use of anti-coagulants (coumadin, heparin, aspirin >325 mg per day).
* Use of any investigational drug within the past 30 days
* Inflammatory arthritis (e.g., rheumatoid or psoriatic arthritis)
* Currently participating in another intervention research study
* Unwilling to be randomized
* Plan to move residence away from the immediate area within the next 2 months
* Drug or alcohol abuse sufficient to hinder compliance with treatment or follow-up procedures
* Pregnant or lactating
* Exclusive use of a wheel chair
* Surgery in either knee in past one year

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2007-04; Primary Completion 2010-04 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian M. Berman, MD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland Center for Integrative Medicine Kernan Hospital, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Lao L, Hochberg M, Lee DYW, Gilpin AMK, Fong HHS, Langenberg P, Chen K, Li EK, Tam LS, Berman B. Huo-Luo-Xiao-Ling (HLXL)-Dan, a Traditional Chinese Medicine, for patients with osteoarthritis of the knee: a multi-site, randomized, double-blind, placebo-controlled phase II clinical trial. Osteoarthritis Cartilage. 2015 Dec;23(12):2102-2108. doi: 10.1016/j.joca.2015.06.007. Epub 2015 Jun 20. PMID 26099553

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began in April 2007 and ended June 2011.
Pre-assignment Details: 2-week run-in period of intermediate-dose: 4,000 mg HLXL If no serious adverse events reported after 2 weeks, the high dose (5,600 mg/day) given for 6 additional weeks.
  Placebo: 14 #0 size gelatin capsules per day, orally, for 8 weeks. Intermediate-dose placebo (2-week run-in) (10 capsules daily) Highest-dose placebo (14 capsules daily)
Groups:
- HLXL: Active herb
  HLXL: Three daily dosages will be investigated. The lowest dosage condition will be 6 capsules (2,400 mg) daily, followed by an escalation to the 10 capsule condition (4,000 mg), and then to the 14 capsule (5,600 mg) condition. Participants will be treated for 6 weeks
- Placebo: Placebo
  The placebo was made from a list of FDA approved ingredients/excipient that matched the color and taste of the real HLXL herbal extract, instead of just white powder used in other placebo trials. Same size and color of capsules were used for the placebo and herbal extract. The equivalent number of capsules used in the treatment group at each dose level were administered to patients assigned to the control group.
Period: Overall Study
Arm/Group | HLXL | Placebo
Started | 47 | 45
Completed | 45 | 42
Not Completed | 2 | 3
Not completed — Lost to Follow-up | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- HLXL: Active herb
  HLXL: Two daily dosages will be investigated. The lowest dosage condition will be 10 capsules (4000 mg) daily for the first two weeks to evaluate safety, followed by an escalation to the 14 capsule condition (5,600 mg). Participants will be treated for 8 weeks.
- Placebo: Placebo
  Placebo: Subjects in the placebo group received an equal number of placebo capsule.
- Total: Total of all reporting groups
Arm/Group | HLXL | Placebo | Total
Number analyzed (Participants) | 47 | 45 | 92
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (9) | 60 (9) | 60 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 32 | 64
  Male | 15 | 13 | 28

OUTCOME MEASURES:

1. Primary Outcome: ‡Pain Normalized Score
Description: ‡Pain normalized score and function normalized score are on a scale of 0-10, with 10 indicating extreme pain/difficulty related to knee arthritis and 0 indicating no pain/difficultly related to knee arthritis.
Time Frame: 8 weeks
Population: Same as baseline.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- HLXL: Active herb
  HLXL: Two daily dosages will be investigated. The subjects in the HLXL group received the medium dose of HLXL (10 capsules/day or 4,000mg/day) in the first 2 weeks to evaluate safety. If no adverse effects were observed, the dose was increased to 14 capsules per day (5,600 mg/day) for the subsequent 6 weeks.
- Placebo: Placebo HLXL
  Placebo: Subjects in the placebo group received an equal number of placebo capsule.
Arm/Group | HLXL | Placebo
Number analyzed (Participants) | 47 | 45
Units on a scale | 3.3 (1.9) | 2.7 (1.7)
Statistical Analysis 1: Comparison: HLXL vs Placebo; Test type: Superiority; p = 0.05, t-test, 2 sided

2. Secondary Outcome: Function Normalized Score
Description: Pain normalized score and function normalized score are on a scale of 0-10, with 10 indicating extreme pain/difficulty related to knee arthritis and 0 indicating no pain/difficultly related to knee arthritis. Overall normalized score is on a scale of 0-30, and is the sum of the pain, stiffness and function normalized scores (each on a scale of 0-10).
Time Frame: 8-Weeks
Population: Same as baseline.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Placebo: Placebo HLXL
  HLXL: Subjects in the placebo group received an equal number of placebo capsule.
Arm/Group | HLXL | Placebo
Number analyzed (Participants) | 46 | 44
Units on a scale | 3.6 (2.0) | 2.7 (1.4)

3. Secondary Outcome: Patient Global Assessment
Description: §Patient Global Assessment is on a scale of 1-5, with 5 indicating excellent and 1 indicating poor (in response to the question "Considering all the ways that your osteoarthritis of the knee affects you, how are you feeling today?")
Time Frame: 8 weeks
Population: Same as baseline
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | HLXL | Placebo
Number analyzed (Participants) | 47 | 45
Units on a scale | 2.7 (1.0) | 2.7 (1.0)

ADVERSE EVENTS:
Time Frame: 8-weeks
Groups:
- HLXL: Active herb
  HLXL: Two daily dosages will be investigated. The subjects in the HLXL group received the medium dose of HLXL (10 capsules/day or 4,000mg/day) in the first 2 weeks to evaluate safety. If no adverse effects were observed, the dose was increased to 14 capsules per day (5,600 mg/ day) for the subsequent 6 weeks.
- Placebo: Placebo HLXL
  Subjects in the placebo group received an equal number of placebo capsule.
Arm/Group | HLXL | Placebo
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/45
Other Adverse Events (participants affected / at risk) | 5/47 | 5/45
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HLXL (N=47) | Placebo (N=45)
GI complaint (General disorders) | 5 (7) | 5 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No